CLINICAL TRIAL: NCT06320587
Title: Determination of the Effect of Kangaroo Care Applied to Premature Newborns by Their Parents on the Newborn's Vital Signs, Parents' Perceived Parenting Self-Efficacy Level and Infant Attachment
Brief Title: The Effect of Kangaroo Care on Parents' Perceived Parenting Self-Efficacy, Infant Attachment and Newborn Vital Signs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: AEŞH-EK1-2023-508
Record Dates: First submitted 2024-02-12; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Kangaroo Care; Fathers; Mother-Infant Interaction; Premature Infant
Keywords: kangaroo care
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Newborns in this group will be given kangaroo care by both their mother and father.
  Interventions: Other: Kangaroo care practice by both mother and father
- Control group (Placebo Comparator): Newborns in this group will be given kangaroo care by only the mother.
  Interventions: Other: Kangaroo care practice only mother

INTERVENTIONS:
Other: Kangaroo care practice by both mother and father — In this group, kangaroo care will be done by both mother and father. Mothers used the Mother-Infant Attachment Scale and the Perceived Maternal Parenting Self-Efficacy Scale as pretests; Fathers will also complete the Postpartum Father-Infant Attachment Survey and the Perceived Father Parenting Self-Efficacy Form. Mothers and fathers in the application group will be provided with kangaroo care for 45 minutes, 2 days a week for 5 weeks. The baby's vital signs will be monitored 30 minutes before each kangaroo care, at the 15th minute of each kangaroo care, and 30 minutes after the kangaroo care, and will be recorded on the Kangaroo Care Monitoring Form. After kangaroo care was completed at the end of 5 weeks, mothers used the Mother-Baby Attachment Scale and the Perceived Mother Parenting Self-Efficacy Scale as posttests; Postnatal Father-Infant Attachment Questionnaire and Perceived Father Parenting Self-Efficacy Form will be filled out by fathers.
  Arms: Experimental group
Other: Kangaroo care practice only mother — In the control group, only the mother will care for the kangaroo. The application will be similar to the experimental group.
  Arms: Control group

SUMMARY:
This study was planned to determine the effect of kangaroo care applied by parents of premature newborns in the neonatal intensive care unit on the newborn's vital signs, perceived parenting self-efficacy level and attachment to the baby.

DETAILED DESCRIPTION:
The research is a randomized controlled trial and an experimental research design will be used. The research will be carried out with two groups as experimental (newborns given kangaroo care by both mother and father) and control (newborns given kangaroo care only by the mother) groups.

ELIGIBILITY:
Inclusion Criteria:

* Parents who volunteered to participate in the research
* Parents who are Turkish citizens and speak Turkish
* Preterm baby born between 28-37 weeks staying in the neonatal intensive care unit
* The mother and father do not have any obstacles in taking care of the kangaroo.
* Mothers and fathers who can come to the hospital regularly on the specified days will be included in the study.

Exclusion Criteria:

* Not volunteering to participate in the research
* Parent's inability to speak Turkish
* Presence of a life-threatening major malformation or serious perinatal complication in the premature baby
* Babies with umbilical catheters and central venous catheters will not be included in the study.

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Mother-To-Infant Bonding Scale | It is designed to be applied from the first day after birth. It will be filled in before kangaroo care and after 5 weeks of kangaroo care.
  It will be applied to evaluate the mother's attachment level to her baby. The lowest score that can be obtained from the scale is 0 and the highest score is 24. The higher the score from the scale, the more it indicates a mother-infant attachment problem.
Perceived Mother Parenting Self-Efficacy Scale | It will be filled in before kangaroo care and after 5 weeks of kangaroo care.
  It will be applied to measure mothers' perceived parenting self-efficacy. The scale consists of 3 sub-dimensions. These; care procedures, the belief in developing positive baby behaviors, the belief in recognizing the baby's behavior, and mother-baby interaction. The lowest score that can be obtained from the scale is 18 and the highest score is 72.As the score obtained increases, the degree of self-efficacy in mothers increases.
Postnatal Paternal-Infant Attachment Questionnaire | It will be filled in before kangaroo care and after 5 weeks of kangaroo care.
  It will be applied to measure fathers' attachment levels to their babies. The lowest score that can be obtained from the scale is 18 and the highest score is 90.A high score from the scale indicates high bonding.
Perceived Father Parenting Self-Efficacy Form | It will be filled in before kangaroo care and after 5 weeks of kangaroo care.
  It is aimed to determine the change in fathers' perceived parenting self-efficacy levels. The lowest score that can be obtained from the form is 0 and the highest score is 10. As the score increases, the degree of self effiacy in father increases.
Physiological parameters of the premature infant: peak heart rate (BPM) | Change from baseline at 5 weeks.
  It shows heart rate per minute of the infant. The normal peak heart rate should be between 100-160 BPM.
Physiological parameters of the premature infant: oxygen saturation (%) | Change from baseline at 5 weeks.
  Oxygen saturation measures the percentage of oxyhemoglobin in the blood. The normal oxygen saturation should be between % 88 - % 100.
Physiological parameters of the premature infant: body temperature (°C) | Change from baseline at 5 weeks.
  It shows body temperature of the infant. The normal body temperature of premature babies should be between 36,5 °C and 37,4 °C.
Physiological parameters of the premature infant:Respiration rate (RPM) | Change from baseline at 5 weeks.
  It shows respiratory rate per minute of the infants. The normal respiratory rate of premature babies should be in the range of 40-60 RPM.

CONTACTS AND LOCATIONS:
Overall Officials: Gönül Kurt, Assoc.Prof, Principal Investigator — Gülhane Sağlık Bilimleri University
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)